CLINICAL TRIAL: NCT07348081
Title: Real World Evidence to Assess the Value of a Digital Care Coordination and Monitoring Program for Supporting Caregivers of Adults Discharged From the Emergency Department.
Acronym: RW-HOMECARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Monka Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 782_RW-HOMECARE; ID RCB : 2025-A02182-47 (Other: ANSM)
Record Dates: First submitted 2025-12-11; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Frailty Syndrome; Caregiver Burden for Those Who Care for Adults With Impaired Functional Status
Keywords: Frailty syndrome; Non-professional caregiver; Burden
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: This is a prospective, longitudinal, single-center pilot study designed to evaluate the effects of the proposed use of the Monka digital solution in real-world conditions and in accordance with the principles of VBHC (Value-Based Health Care), a systemic approach aimed at maximizing the value of care for patients, defined as the ratio between the clinical results obtained and the resources mobilized to achieve them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient and caregiver dyad experiencing the MyMonka solution in real-life conditions (Experimental)
  Interventions: Other: Caregivers supporting vulnerable patients and using the MyMonka solution.

INTERVENTIONS:
Other: Caregivers supporting vulnerable patients and using the MyMonka solution. — Testing of the MyMonka solution; Response to questionnaires during the follow-up period on quality of life and burden measurement

SUMMARY:
The RW-HOMECARE study is a prospective, longitudinal, real-world pilot trial designed to assess the impact of proposing the Monka digital solution to non-professional caregivers of patients discharged from emergency or short-stay units. The primary objective is to measure changes in caregiver burden using the ZBI-12 scale at baseline, 30 days, and 90 days. Secondary objectives include evaluating caregivers' physical and mental quality of life (SF-12), patient frailty (Clinical Frailty Scale), and the incidence of adverse events such as emergency visits, unplanned hospitalizations, falls, institutionalization, and death within 90 days. The study also examines the usability, acceptability, and satisfaction with Monka digital solution through standardized questionnaires, the correlation between algorithm-generated vulnerability scores and established measures, and reasons for non-adoption.

Eligible dyads (patient and caregiver) are recruited at discharge from emergency or short-stay units. After informed consent, caregivers receive free access to Monka digital solution for 3 months, along with a user guide. Follow-up assessments are conducted by phone at Day 30 and Day 90 (±14 days). All interventions by the coordinating nurse are tracked and analyzed quantitatively and qualitatively.

ELIGIBILITY:
Inclusion Criteria:

FOR THE PATIENT

* Person aged 18 or over, treated in the Emergency Department or Emergency Beds
* Affiliated with Social Security
* Having an adult non-professional relative helping them with one or more activities of daily living
* Having a medical decision to return home within the next 72 hours
* Who has given their free, informed, and express consent FOR THE CAREGIVER
* Individuals aged 18 or older
* Who are non-professional caregivers as defined in Article L. 113-1-3 of the Social Action and Families Code, living with or separately from the person being cared for (20)
* Providing assistance to the patient with one or more activities of daily living, i.e., shopping, medical appointments, coordination of care, administrative tasks, and moral support
* Access to a cell phone, computer, or tablet with an internet connection
* Having given their free, informed, and express consent

Exclusion Criteria:

FOR THE PATIENT

* Non-French speakers
* People living in a medical institution or scheduled for institutionalization within the next 3 months
* People receiving home hospitalization (HAD) or palliative care at home
* People under legal protection, deprived of their liberty, or under legal guardianship (tutelage or curatelle) FOR THE CAREGIVER
* Non-French speakers
* People with cognitive or psychiatric disorders that prevent them from understanding and using the MONKA solution
* People under legal protection, deprived of their liberty, or under legal guardianship (tutelage or curatelle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Change in the score on the 12-item Zarit Burden Interview questionnaire (ZBI-12, Appendix 1), measured on days 0, 30, and 90, among family caregivers participating in the study. | Days 0, 30 and 90

SECONDARY OUTCOMES:
Change in the physical and mental quality of life of caregivers, expressed as the difference between SF-12 questionnaire scores at baseline, on day 30, and on day 90. | Days 30 and 90
Change in patient frailty expressed as the difference between the Clinical Frailty Scale score obtained at inclusion and on day 90. | Days 0 and 90
Percentage of people affected by the following adverse events within three months of returning home: new emergency room visits, unscheduled hospitalizations and their duration, falls, home hospitalizations, institutionalization, and death. | Days 90
Evaluation of the use, acceptability, usability, and impact of the Monka digital solution for caregivers through intervention tracking, algorithm-based vulnerability assessment, and standardized questionnaires over a 90-day period. | Days 0 and 90

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided